CLINICAL TRIAL: NCT06465329
Title: A Randomized Phase 2 Platform Study to Evaluate Cemiplimab Plus Chemotherapy Versus Cemiplimab Plus Chemotherapy Plus Other Cancer Treatments for the Perioperative Treatment of Patients With Resectable Non-Small Cell Lung Cancer
Brief Title: A Study of Cemiplimab Plus Chemotherapy Versus Cemiplimab Plus Chemotherapy Plus Other Cancer Treatments for Adult Patients With Operable Non-Small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-2268; 2023-509806-31-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Carcinoma; Resectable NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — cemiplimab; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemotherapy+Cemiplimab (Active Comparator): Control treatment
  Interventions: Drug: Cemiplimab; Drug: Platinum-based chemotherapy
- Arm 1: Chemotherapy+Cemiplimab+REGN7075 (Experimental): Investigational Treatment
  Interventions: Drug: Cemiplimab; Drug: Platinum-based chemotherapy; Drug: REGN7075

INTERVENTIONS:
Drug: Cemiplimab — Intravenous (IV) infusion administration
  Other Names: REGN2810; LIBTAYO
Drug: Platinum-based chemotherapy — IV infusion
Drug: REGN7075 — IV infusion
  Other Names: EGFRxCD28 bispecific immunotherapy
  Arms: Arm 1: Chemotherapy+Cemiplimab+REGN7075

SUMMARY:
This study will enroll adult participants with early-stage (stage II-IIIB) non-small cell lung cancer for whom surgery is planned.

The aim is to find out whether an investigational treatment (consisting of the immunotherapy drug cemiplimab plus chemotherapy plus a third drug) works better than cemiplimab plus chemotherapy without the additional drug.

The study is also looking at several other research questions, including:

* What are the side effects associated with the investigational treatments in comparison to the control treatment?
* Do the investigational treatments or the control treatment have an effect on the type of surgery that is performed?
* How much of the study drug(s) are in the blood at a given time?
* Does the body make antibodies against the study drug(s) (which could make the drug(s) less effective or could lead to side effects)?

ELIGIBILITY:
General Key Inclusion Criteria:

1. Histologically confirmed stage II through IIIB (N2) NSCLC, that is considered resectable with curative intent, as described in the protocol
2. Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1
3. Available formalin-fixed paraffin-embedded (FFPE) tumor sample blocks for submission, as described in the protocol
4. Eastern Cooperative Oncology Group Performance Status scale (ECOG PS) of 0 to 1
5. Adequate organ and bone marrow function, as described in the protocol

General Key Exclusion Criteria:

1. Any systemic anti-cancer therapy or radiotherapy for the current tumor, as described in the protocol
2. Presence of known oncogenic alterations in epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) in the tumor prior to randomization, as described in the protocol
3. Presence of grade≥ 2 peripheral neuropathy
4. Another malignancy that is progressing or requires active treatment, as described in the protocol

Arm Specific Exclusion Criteria:

Arm 1:

1. Grade ≥3 hypercalcemia, as defined in the protocol
2. Any central nervous system (CNS) pathology that could increase the risk of immune effector cell-associated neurotoxicity syndrome (ICANS), as described in the protocol
3. Has marked baseline prolongation of the time from the start of the Q wave to the end of the T wave in electrocardiogram (QT)/corrected QT interval (QTc) interval or risk factors for prolonged QTc, as described in the protocol

Note: Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2030-05-02 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) rate as determined by central blinded independent pathology review (BIPR) | Up to 12 weeks

SECONDARY OUTCOMES:
Pathologic complete response (pCR) rate as determined by central BIPR | Up to 12 weeks
Residual viable tumor (RVT) as determined by central BIPR | Up to 12 weeks
Median event-free survival (EFS) | Up to 5 years
EFS rate | Up to 5 years
Objective response rate (ORR) | Up to 9 weeks
Overall survival (OS) | Up to 5 years
Incidence of treatment-emergent adverse events (TEAEs) | Up to 76 weeks
Severity of TEAEs | Up to 76 weeks
Incidence of TEAEs leading to death | Up to 76 weeks
Incidence of TEAEs leading to treatment discontinuation | Up to 76 weeks
Incidence of serious adverse events (SAEs) | Up to 76 weeks
Incidence of adverse events of special interest (AESIs) | Up to 76 weeks
Incidence of immune-mediated adverse events (imAEs) | Up to 76 weeks
Incidence of infusion-related reactions (IRRs) | Up to 76 weeks
Incidence of grade ≥3 laboratory abnormalities | Up to 76 weeks
  As assessed by the Common Terminology Criteria for Adverse Events (CTCAE) grading system version 5.0 (for all grades)
Proportion of delayed surgeries due to TEAEs | Up to 76 weeks
Proportion of cancelled surgeries due to TEAEs | Up to 76 weeks
Incidence of anti-drug antibodies (ADAs) to cemiplimab over time | Up to 67 weeks
Titer of ADAs to cemiplimab over time | Up to 67 weeks
Incidence of ADAs to novel anti-cancer agents over time | Up to 67 weeks
Titer of ADAs to novel anti-cancer agents over time | Up to 67 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (49):
- United States (14):
  - University of California Irvine, Orange, California
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Providence Portland Medical Center, Portland, Oregon
  - University Of Nebraska Medical Center, Portland, Oregon
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Prairie Lakes Healthcare System, Watertown, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute (SCRI) Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - BRCC/Oncology & Hematology Associates of SW Virginia, Blacksburg, Virginia
- Brazil (11):
  - Oncology Clinical Research Center, Cachoeiro de Itapemirim, Espírito Santo
  - Instituto Mario Penna, Belo Horizonte, Minas Gerais
  - Instituto Sul Mineiro De Oncologia LTDA, Pouso Alegre, Minas Gerais
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco
  - Liga Norte Riograndense Contra o Cancer, Natal, Rio Grande do Norte
  - Hospital Mae de Deus Integrated Oncology Center, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Ynova Pesquisa Clinica, Florianópolis, Santa Catarina
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Unimed Sorocaba, Sorocaba, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
- France (7):
  - CHU Rennes, Rennes, Brittany Region
  - Centre Hospitalier Intercommunal Toulon - CHITS, Toulon, Var
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Clinique Belharra, Bayonne
  - CHU Grenoble Alpes, Grenoble
  - Montpellier Academic Hospital, Montpellier
  - Institut Curie, Paris, Île-de-France Region
- Germany (4):
  - Klinikum Kassel GmbH, Hauttumorzentrum, Kassel, Hesse
  - University Medicine Gottingen, Göttingen, Lower Saxony
  - University of Leipzig, Leipzig, Saxony
  - University Hospital RWTH Aachen, Aachen
- Spain (12):
  - Catalan Instituye of Oncology Badalona, Badalona, Barcelona
  - Hospital Valdecilla, Santander, Cantabria
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Virgen del Rocio, Seville
  - Hospital Clinico Universitario Valencia, Valencia
  - Consorci Hospital General Universitario de Valencia, Valencia
  - Hospital Clinico Lozano Blesa, Zaragoza
- Florya Medical Park Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/